CLINICAL TRIAL: NCT06273384
Title: Diagnostic Performance of Current Infection Marker (CIM) for Helicobacter Pylori Infection in Patients With Peptic Ulcer Bleeding
Brief Title: Diagnostic Performance of CIM for Helicobacter Pylori Infection in Patients With Peptic Ulcer Bleeding
Acronym: CIM
Status: Not yet recruiting | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Watcharasak Chotiyaputta, Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Thailand, Mahidol University
Other Study IDs: Si 062/2023
Record Dates: First submitted 2024-02-07; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Helicobacter Pylori Infection; Peptic Ulcer Hemorrhage
Keywords: Helicobacter Pylori Infection; Peptic Ulcer Hemorrhage; Current infection marker
MeSH Terms: conditions — Peptic Ulcer Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Participants underwent esophagogastroduodenoscopy (EGD) with random biopsies of two pieces of gastric mucosa: one from the antrum and another from the incisura angularis. Subsequently, PCR was performed for the detection of H. pylori DNA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention group: Patients aged 18 years and older who present with peptic ulcer hemorrhage, confirmed by esophagogastroduodenoscopy (EGD).

SUMMARY:
The goal of this cross-sectional study is to evaluate the efficacy of current infection marker (CIM) method for H. pylori detection. The main questions it aims to answer are:

* To evaluate the efficacy of CIM method for H. pylori detection compared to rapid urease test(RUT), histopathology, polymerase chain reaction (PCR), and urea breath test (UBT) in patients who presented with upper gastrointestinal hemorrhage from peptic ulcer, and their sensitivity, specificity, accuracy, positive predictive value (PPV), negative predictive value (NPV), positive likelihood ratio, and negative likelihood ratio.
* To evaluate the advantages of CIM method for H. pylori detection comparing to RUT, histopathology, PCR, and UBT in patients who presented with upper gastrointestinal hemorrhage from peptic ulcer as net reclassification index (NRI).
* To study the associated factors in false negative value of H. pylori detection methods with CIM, RUT, histopathology, PCR, and UBT.

DETAILED DESCRIPTION:
Helicobacter pylori (H. pylori) is a Gram-negative bacillus that involves gastric mucosa and was first isolated in 1982. The global prevalence of H. pylori infection is about 50% and the prevalence is different in each region of the world. The highest prevalence of H. pylori infection is up to 70.1% in Africa, but the prevalence in the South-East Asian region varies from 28.6 to 70.3%. For Thailand, the prevalence of H. pylori infection was reported approximately 43.6-64.0%. H. pylori infection is also well-known to be associated with gastric cancer, Gastric mucosa-associated lymphoid tissue (MALT) lymphoma, and peptic ulcer.

Peptic ulcer strongly associates with H. pylori infection. The global prevalence of H. pylori infection is 48.5-94.5% and 66.9-95.8% in gastric ulcer and duodenal ulcer, respectively. These data corresponded to the prevalence in Thailand which is 68.9% and 82.8 % in gastric ulcers and duodenal ulcers, respectively. Peptic ulcer is also one of the common causes of upper gastrointestinal hemorrhage. In contrast, H. pylori eradication has been shown to reduce the risk of recurrent upper gastrointestinal bleeding.

Nowadays, there are several tests for H. pylori infection including endoscopic-based methods such as rapid urease test (RUT), histopathology, culture, and polymerase chain reaction (PCR) for deoxyribonucleic acid (DNA) of H. pylori detection, and non-invasive methods, including urea breath test (UBT), fecal antigen test, and serologic test. In clinical practice, patients under upper gastrointestinal endoscopy with suspicion of H. pylori infection are almost always tested with RUT and histopathology. Both these methods are simple and available with high sensitivity and specificity that is greater 90 and 95%, respectively.

Patients presented with upper gastrointestinal bleeding are recommended to be diagnosed and treated with endoscopy, if the peptic ulcer including gastric ulcer or duodenal ulcer was found, the H. pylori infection must be considered to test. Blood in the gastric cavity, proton pump inhibitor (PPI), and antibiotic prescription can decrease the sensitivity and specificity of RUT and histopathology. Moreover, the patients with gastric ulcer and duodenal ulcer should be generally treated with PPI for a total duration of 8 to 12 weeks and 4 to 8 weeks, respectively, which could affect the accuracy of RUT for H. pylori detection. Although PCR technique has more than 98% of sensitivity, specificity, and accuracy, it is very expensive test that requires high performance center, so PCR test is not always available and not suitable for clinical practice. Therefore, these limitations can delay the diagnosis of H. pylori infection in patients with upper gastrointestinal hemorrhage, so the patients are also not treated this infection in timely manner.

Serology test for H. pylori infection is the test for blood immunoglobulin G (IgG) detection that has 85% sensitivity and 79% specificity 26. PPI or antibiotic uses and upper gastrointestinal bleeding do not affect to this test, so this method might be a better test for H. pylori infection than the endoscopic-based tests including RUT or histopathology. Currently, the immunochromatographic test is a novel method for H. pylori infection that identify current infection marker (CIM) of H. pylori. It is a simple and rapid test in which the sensitivity and the specificity in general population are 90 - 92.3% and 89 - 90.5%, respectively. However, the use of CIM for H. pylori infection in patients with upper gastrointestinal hemorrhage from peptic ulcer who are treated with PPI or antibiotic has not been done yet.

This study aims to evaluate the efficacy of CIM for H. pylori infection test in patients with upper gastrointestinal hemorrhage from peptic ulcer compared to rapid urease test, histopathology, PCR for H. pylori detection, and UBT method.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Upper gastrointestinal hemorrhage and undergo esophagogastroduodenoscopy with diagnosis of peptic ulcer

Exclusion Criteria:

* Inappropriate gastric mucosal biopsy conditions such as hemodynamic instability, coagulopathy or severe thrombocytopenia or massive bloody content in gastric cavity or duodenum
* Previous history of gastric surgery such as partial or total gastrectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years or older, who present with upper gastrointestinal hemorrhage and undergo esophagogastroduodenoscopy, receiving a diagnosis of peptic ulcer, will be recruited and enrolled. The exclusion criteria include patients with inappropriate gastric mucosal biopsy conditions, such as hemodynamic instability, coagulopathy, severe thrombocytopenia, or the presence of massive bloody content in the gastric cavity or duodenum. Additionally, individuals with a previous history of gastric surgery, such as partial or total gastrectomy, will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The efficacy of CIM method for H. pylori detection | Through study completion, an average of 2 years
  The sensitivity, specificity, and accuracy of the CIM method for H. pylori detection were compared to those of RUT, histopathology, PCR, and UBT.

SECONDARY OUTCOMES:
The advantages of CIM method for H. pylori detection | Through study completion, an average of 2 years
  The net reclassification index (NRI) of the CIM method for H. pylori detection were compared to those of RUT, histopathology, PCR, and UBT.

CONTACTS AND LOCATIONS:
Overall Officials: Monthira Maneerattanaporn, Asso Prof, Principal Investigator — Department of Medicine, Siriraj Hospital, Mahidol University, Bangkok, Thailand
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok Noi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Warren JR, Marshall B. Unidentified curved bacilli on gastric epithelium in active chronic gastritis. Lancet. 1983 Jun 4;1(8336):1273-5. No abstract available. PMID 6134060
- [Result] Pounder RE, Ng D. The prevalence of Helicobacter pylori infection in different countries. Aliment Pharmacol Ther. 1995;9 Suppl 2:33-9. PMID 8547526
- [Result] Hooi JKY, Lai WY, Ng WK, Suen MMY, Underwood FE, Tanyingoh D, Malfertheiner P, Graham DY, Wong VWS, Wu JCY, Chan FKL, Sung JJY, Kaplan GG, Ng SC. Global Prevalence of Helicobacter pylori Infection: Systematic Review and Meta-Analysis. Gastroenterology. 2017 Aug;153(2):420-429. doi: 10.1053/j.gastro.2017.04.022. Epub 2017 Apr 27. PMID 28456631
- [Result] Sirinthornpunya S. Prevalence of Helicobacter pylori infection in patients with peptic disease. J Med Assoc Thai. 2012 Mar;95 Suppl 3:S22-7. PMID 22619883
- [Result] Hentschel E, Brandstatter G, Dragosics B, Hirschl AM, Nemec H, Schutze K, Taufer M, Wurzer H. Effect of ranitidine and amoxicillin plus metronidazole on the eradication of Helicobacter pylori and the recurrence of duodenal ulcer. N Engl J Med. 1993 Feb 4;328(5):308-12. doi: 10.1056/NEJM199302043280503. PMID 8419816
- [Result] Moayyedi P. The health economics of Helicobacter pylori infection. Best Pract Res Clin Gastroenterol. 2007;21(2):347-61. doi: 10.1016/j.bpg.2006.11.004. PMID 17382282
- [Result] Ford AC, Moayyedi P. Whom should we "test and treat" for Helicobacter pylori? BMJ. 2014 May 20;348:g3320. doi: 10.1136/bmj.g3320. No abstract available. PMID 24846521
- [Result] McColl KE. Clinical practice. Helicobacter pylori infection. N Engl J Med. 2010 Apr 29;362(17):1597-604. doi: 10.1056/NEJMcp1001110. No abstract available. PMID 20427808
- [Result] Ciociola AA, McSorley DJ, Turner K, Sykes D, Palmer JB. Helicobacter pylori infection rates in duodenal ulcer patients in the United States may be lower than previously estimated. Am J Gastroenterol. 1999 Jul;94(7):1834-40. doi: 10.1111/j.1572-0241.1999.01214.x. PMID 10406244
- [Result] Tsuji H, Kohli Y, Fukumitsu S, Morita K, Kaneko H, Ohkawara T, Minami M, Ueda K, Sawa Y, Matsuzaki H, Morinaga O, Ohkawara Y. Helicobacter pylori-negative gastric and duodenal ulcers. J Gastroenterol. 1999 Aug;34(4):455-60. doi: 10.1007/s005350050296. PMID 10452677
- [Result] Vu C, Ng YY. Prevalence of Helicobacter pylori in peptic ulcer disease in a Singapore hospital. Singapore Med J. 2000 Oct;41(10):478-81. PMID 11281437
- [Result] Zhang W, Liang X, Chen X, Ge Z, Lu H. Time trends in the prevalence of Helicobacter pylori infection in patients with peptic ulcer disease: a single-center retrospective study in Shanghai. J Int Med Res. 2021 Oct;49(10):3000605211051167. doi: 10.1177/03000605211051167. PMID 34686094
- [Result] Lanas A, Chan FKL. Peptic ulcer disease. Lancet. 2017 Aug 5;390(10094):613-624. doi: 10.1016/S0140-6736(16)32404-7. Epub 2017 Feb 25. PMID 28242110
- [Result] Jaspersen D, Koerner T, Schorr W, Brennenstuhl M, Raschka C, Hammar CH. Helicobacter pylori eradication reduces the rate of rebleeding in ulcer hemorrhage. Gastrointest Endosc. 1995 Jan;41(1):5-7. doi: 10.1016/s0016-5107(95)70267-9. PMID 7698624
- [Result] Rokkas T, Karameris A, Mavrogeorgis A, Rallis E, Giannikos N. Eradication of Helicobacter pylori reduces the possibility of rebleeding in peptic ulcer disease. Gastrointest Endosc. 1995 Jan;41(1):1-4. doi: 10.1016/s0016-5107(95)70266-0. PMID 7698617
- [Result] FitzGerald R, Smith SM. An Overview of Helicobacter pylori Infection. Methods Mol Biol. 2021;2283:1-14. doi: 10.1007/978-1-0716-1302-3_1. PMID 33765303
- [Result] Patel SK, Pratap CB, Jain AK, Gulati AK, Nath G. Diagnosis of Helicobacter pylori: what should be the gold standard? World J Gastroenterol. 2014 Sep 28;20(36):12847-59. doi: 10.3748/wjg.v20.i36.12847. PMID 25278682
- [Result] Chey WD, Wong BC; Practice Parameters Committee of the American College of Gastroenterology. American College of Gastroenterology guideline on the management of Helicobacter pylori infection. Am J Gastroenterol. 2007 Aug;102(8):1808-25. doi: 10.1111/j.1572-0241.2007.01393.x. Epub 2007 Jun 29. PMID 17608775
- [Result] Gralnek IM, Dumonceau JM, Kuipers EJ, Lanas A, Sanders DS, Kurien M, Rotondano G, Hucl T, Dinis-Ribeiro M, Marmo R, Racz I, Arezzo A, Hoffmann RT, Lesur G, de Franchis R, Aabakken L, Veitch A, Radaelli F, Salgueiro P, Cardoso R, Maia L, Zullo A, Cipolletta L, Hassan C. Diagnosis and management of nonvariceal upper gastrointestinal hemorrhage: European Society of Gastrointestinal Endoscopy (ESGE) Guideline. Endoscopy. 2015 Oct;47(10):a1-46. doi: 10.1055/s-0034-1393172. Epub 2015 Sep 29. PMID 26417980
- [Result] Laine L, Barkun AN, Saltzman JR, Martel M, Leontiadis GI. ACG Clinical Guideline: Upper Gastrointestinal and Ulcer Bleeding. Am J Gastroenterol. 2021 May 1;116(5):899-917. doi: 10.14309/ajg.0000000000001245. PMID 33929377
- [Result] Lee JM, Breslin NP, Fallon C, O'Morain CA. Rapid urease tests lack sensitivity in Helicobacter pylori diagnosis when peptic ulcer disease presents with bleeding. Am J Gastroenterol. 2000 May;95(5):1166-70. doi: 10.1111/j.1572-0241.2000.02004.x. PMID 10811322
- [Result] Gatta L, Vakil N, Ricci C, Osborn JF, Tampieri A, Perna F, Miglioli M, Vaira D. Effect of proton pump inhibitors and antacid therapy on 13C urea breath tests and stool test for Helicobacter pylori infection. Am J Gastroenterol. 2004 May;99(5):823-9. doi: 10.1111/j.1572-0241.2004.30162.x. PMID 15128344
- [Result] Gisbert JP, Abraira V. Accuracy of Helicobacter pylori diagnostic tests in patients with bleeding peptic ulcer: a systematic review and meta-analysis. Am J Gastroenterol. 2006 Apr;101(4):848-63. doi: 10.1111/j.1572-0241.2006.00528.x. Epub 2006 Feb 22. PMID 16494583
- [Result] Singh V, Mishra S, Rao GR, Jain AK, Dixit VK, Gulati AK, Mahajan D, McClelland M, Nath G. Evaluation of nested PCR in detection of Helicobacter pylori targeting a highly conserved gene: HSP60. Helicobacter. 2008 Feb;13(1):30-4. doi: 10.1111/j.1523-5378.2008.00573.x. PMID 18205663
- [Result] Jehanne Q, Benejat L, Megraud F, Bessede E, Lehours P. Evaluation of the Allplex H pylori and ClariR PCR Assay for Helicobacter pylori detection on gastric biopsies. Helicobacter. 2020 Aug;25(4):e12702. doi: 10.1111/hel.12702. Epub 2020 May 19. PMID 32426894
- [Result] Loy CT, Irwig LM, Katelaris PH, Talley NJ. Do commercial serological kits for Helicobacter pylori infection differ in accuracy? A meta-analysis. Am J Gastroenterol. 1996 Jun;91(6):1138-44. PMID 8651160
- [Result] Mohammadian T, Ganji L. The Diagnostic Tests for Detection of Helicobacter pylori Infection. Monoclon Antib Immunodiagn Immunother. 2019 Feb;38(1):1-7. doi: 10.1089/mab.2018.0032. Epub 2019 Jan 16. PMID 30648911
- [Result] Rahman SH, Azam MG, Rahman MA, Arfin MS, Alam MM, Bhuiyan TM, Ahmed N, Rahman M, Nahar S, Hassan MS. Non-invasive diagnosis of H pylori infection: evaluation of serological tests with and without current infection marker CIM. World J Gastroenterol. 2008 Feb 28;14(8):1231-6. doi: 10.3748/wjg.14.1231. PMID 18300349
- [Result] Wang XY, Yang Y, Shi RH, Ho B, Wang HD, Zhang GX. An evaluation of a serologic test with a current infection marker of Helicobacter pylori before and after eradication therapy in Chinese. Helicobacter. 2008 Feb;13(1):49-55. doi: 10.1111/j.1523-5378.2008.00578.x. PMID 18205666
- [Result] Forrest JA, Finlayson ND, Shearman DJ. Endoscopy in gastrointestinal bleeding. Lancet. 1974 Aug 17;2(7877):394-7. doi: 10.1016/s0140-6736(74)91770-x. No abstract available. PMID 4136718
- [Result] Gralnek IM, Barkun AN, Bardou M. Management of acute bleeding from a peptic ulcer. N Engl J Med. 2008 Aug 28;359(9):928-37. doi: 10.1056/NEJMra0706113. No abstract available. PMID 18753649
- [Result] Banks M, Graham D, Jansen M, Gotoda T, Coda S, di Pietro M, Uedo N, Bhandari P, Pritchard DM, Kuipers EJ, Rodriguez-Justo M, Novelli MR, Ragunath K, Shepherd N, Dinis-Ribeiro M. British Society of Gastroenterology guidelines on the diagnosis and management of patients at risk of gastric adenocarcinoma. Gut. 2019 Sep;68(9):1545-1575. doi: 10.1136/gutjnl-2018-318126. Epub 2019 Jul 5. PMID 31278206